CLINICAL TRIAL: NCT04848415
Title: Diagnostic Performance of Point of Care Ultrasound to Identify Intestinal Obstruction
Acronym: OCCLUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OCCLUS
Record Dates: First submitted 2021-02-15; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Bowel Obstruction
Keywords: Bowel obstruction; Computed tomography; Ultrasound
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Point-of-Care Ultrasound — Patients admitted to the ED with abdominal pain and suspicion of bowel obstruction : realization of a Point-of-Care Ultrasound after clinical exam by the Emergency Physician in charge as a standard of care. Beside usual findings, the investigators will search for signs of bowel obstruction: dilated and incompressible small bowel loop, back-and-forth peristalsis sign. Determination of probability of small bowel obstruction. Realization of a computed tomography in search of small bowel obstruction.

SUMMARY:
As reported in previous studies, Point-of-Care Ultrasound (POCUS) has good performance for the diagnosis of bowel obstruction even when compared with CT. This inexpensive, radiation-free tool is available in a majority of ED. It is performed at the patient's bedside with immediate results. The learning curve allows Emergency Physicians (EP) to perform this exam after a relative brief training period.

The investigators aim to investigate the ability of POCUS performed before CT to exclude the diagnosis of bowel obstruction in patients admitted for abdominal pain.

DETAILED DESCRIPTION:
Bowel obstruction (BO) is frequently suspected in the Emergency Department (ED). Computed Tomography (CT) is commonly used to diagnose this disease. However, CT is not always available in real-time, requires technician times, is associated with increased cost and exposes patients to radiations.

The researchers will investigate the diagnosis performances of POCUS for the diagnosis of BO with comparison with CT which will be considered as the gold standard. The wain objective will be the ability to exclude the diagnosis of BO, the main criteria being the negative predictive value. The secondary objectives will be the diagnosis performances (sensitivity, specificity, positive predictive value), duration and difficulty of POCUS

ELIGIBILITY:
Inclusion Criteria :

* Adult patients
* Abdominal pain
* Suspected bowel obstruction

Exclusion Criteria :

- Documented end-of-life precluding CT realization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ED for abdominal pain and suspicion of bowel obstruction
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of POCUS | Through ED stay, up to 24 hours
  Negative predictive value of POCUS for the diagnosis of bowel obstruction compared with computed tomography result

SECONDARY OUTCOMES:
Positive predictive value of POCUS for the diagnosis of bowel obstruction | Through ED stay, up to 24 hours
  Positive predictive value
Sensitivity of POCUS for the diagnosis of bowel obstruction | Through ED stay, up to 24 hours
  sensitivity of POCUS, for the diagnosis of bowel obstruction compared with computed tomography result
Specificity of POCUS for the diagnosis of bowel obstruction | Through ED stay, up to 24 hours
  specificity of POCUS, for the diagnosis of bowel obstruction compared with computed tomography result

IPD SHARING:
Plan to Share IPD: No